CLINICAL TRIAL: NCT05054478
Title: Primary Plasma Cell Leukemia: a Prospective Phase 2 Study Incorporating Daratumumab to Chemotherapy and Stem Cell Transplantation : PCL-2 Study
Brief Title: Primary Plasma Cell Leukemia: a Prospective Phase 2 Study Incorporating Daratumumab to Chemotherapy and Stem Cell Transplantation
Acronym: PCL-2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP190205; 2019-004170-26 (EudraCT Number)
Record Dates: First submitted 2021-07-31; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-05

CONDITIONS: Plasma Cell Leukemia
MeSH Terms: conditions — Leukemia, Plasma Cell | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Single-arm phase 2 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): 4 days of dexamethasone. According to local practice, one dose of doxorubicine (30 mg/m2 IV) or cyclophosphamide (750 mg/m2 IV) may also be added
  Induction Treatment (4 months): Subject will receive 4 x 28 days cycles of Dara-VRD induction:
  Daratumumab sc 1800 mg on D1 D8 D15 D22 for cycle1 & 2 and D1 D15 for cycle 3 & 4 Bortezomib sc 1.3 mg/m2 on D1 D4 D8 D11 for each cycle Lenalidomide po 25 mg on D1 to D21 for each cycle Dexamethasone po 20 mg on D1 D2 D8 D9 D15 D16 D22 D23 for each cycle
  High dose melphalan 200mg/m2 as conditioning therapy and first ASCT
  First consolidation : 2 cycles of Dara-VRd
  * Daratumumab 1800 mg s.c D1 D15
  * Bortezomib 1.3 mg/m2 s.c D1 D8 D15 D22
  * Lenalidomide 25 mg p.o from D1 to D21
  * Dexa 20 mg p.o D1 D8 D15 D22
  High dose melphalan 200mg/m2 as conditioning therapy and second ASCT Second consolidation : 6 cycles of Dara-VRd (every 2 months for 2 years) Then maintenance: Lenalidomide every 28 days (25 mg from D1 to D21) for 1 year
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab added to induction, first consolidation and second consolidation

SUMMARY:
Single-Arm phase 2 trial evaluating efficacy of incorporating Daratumumab to treatment of newly diagnosed primary plasma cell leukemia. Treatment will be based on Dara-VRd induction followed by first ASCT, Dara-VRd for first consolidation, second ASCT, Dara-VRd for 1 year as second consolidation and Lenalidomide for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 to 69 years old.
2. Patient with primary plasma cell leukemia disease as defined by the International Myeloma Working Group -IMWG (Annexe I)
3. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
4. Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2.
5. Eligible for high dose Melphalan therapy with ASCT
6. Total bilirubin <= 2 X the upper limit of the normal range (ULN).
7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3 ULN.
8. Calculated creatinine clearance >= 20 mL/min
9. Female patients who:

   * Have been postmenopausal for at least 2 years before the screening visit, OR
   * are surgically sterile, OR If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal and post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
10. Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal and post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
11. Patients agree

    * not to share study medication with any other person and to return all unused study drugs to the investigator.
    * to abstain from donating blood while taking the study drug therapy and for one week following discontinuation of the study drug therapy.
12. Must be able to adhere to the study visit schedule and other protocol requirements
13. Affiliated with an appropriate social security system

Exclusion Criteria:

1. Male or female patients <18 or > 69 years old
2. Prior history of malignancies, unless free of the disease for ≥ 5 years.
3. Prior history of symptomatic myeloma; did not received any previous chemotherapy for myeloma except corticotherapy (dexamethasone 40 mg/d for 4 days max).
4. Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation.
5. Pregnant or breast feeding females
6. Known positive for HIV
7. Known seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as a viremia at least 12 weeks after completion of antiviral therapy)
8. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti- HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
9. Patient with severe renal failure that require dialysis and clearance creatinine < 20 ml/min
10. Prior local irradiation within two weeks before first dose. However, an exception (that is patients allowed to remain in the treatment phase of the study) is made for radiation therapy to a pathological fracture site to enhance bone healing or to treat post-fracture pain that is refractory to narcotic analgesics because pathologic bone fractures do not by themselves fulfil a criterion for disease progression.)
11. Evidence of central nervous system (CNS) involvement
12. Unable to take corticosteroid therapy, daratumumab, bortezomib and or lenalidomide at study entry.
13. Ongoing active infection, especially ongoing pneumonitis
14. Ongoing Cardiac dysfunction: specify e.g. uncontrolled hypertension, MI within 6 months, unstable Angina pectoris, Cardiac arrhythmia Grade 2 or higher, NYHA class III/IV
15. Patients with a left ventricular ejection fraction under to 40 % (LVEF <40%).
16. Use of any other experimental drug or therapy within 15 days of screening.
17. Any >grade 2 toxicity unresolved
18. Inability or unwillingness to comply with birth control requirements
19. Unable to take antithrombotic medicines at study entry
20. Major surgery within 14 days before enrolment
21. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
22. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
23. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of daratumumab and lenalidomide including difficulty swallowing

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
VGPR or better at the completion of induction phase | completion of induction phase [4 Months]
  The VGPR or better rate (as determined by the reviewer) is defined as the proportion of patients with confirmed IMWG criteria for VGPR, CR or stringent CRrelative to the total number of patients in the ITT population

SECONDARY OUTCOMES:
Progression Free Survival | 3 years
Response rates (sCR, CR, VGPR, PR, SD): | after induction [4 months]
Response rates (sCR, CR, VGPR, PR, SD): | after ASCT n°2 [10 months]
Response rates (sCR, CR, VGPR, PR, SD): | after second consolidation phase [22 months]
Response rates (sCR, CR, VGPR, PR, SD): | end of treatment [34 months]
Overall response rate (ORR) | after induction [4 months]
Overall response rate (ORR) | after ASCT n°2 [10 months]
Overall response rate (ORR) | after second consolidation phase [22 months]
Overall response rate (ORR) | end of treatment [34 months]
Overall survival (OS) | 3 years
Time to progression (TTP) | 3 years
Duration of response (DOR) | 3 years
Safety | Whole trial duration [48 months]
  Adverse Events
MRD negative rate assessed by NGS | End of induction [4 months]
MRD negative rate assessed by NGS | after ASCT n°2 [10 months]
MRD negative rate assessed by NGS | after second consolidation phase [22 months]
MRD negative rate assessed by NGS | end of treatment [34 months]
Quality of life | End of induction [4 months]
  defined using EORTC QLQ-C30 domain scores
Quality of life | after ASCT n°2 [10 months]
  defined using EORTC QLQ-C30 domain scores
Quality of life | after second consolidation phase [22 months]
  defined using EORTC QLQ-C30 domain scores

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Royer, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris